CLINICAL TRIAL: NCT06106373
Title: iotaSOFT Insertion System for Use With Cochlear Implant Surgery in Pediatrics
Brief Title: iotaSOFT Pediatric Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iotaMotion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iotaSOFT000002
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral; Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral; Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pediatric Cochlear Implant Recipient (Experimental): Pediatric subjects receiving a cochlear implant between the ages of 9 months and under 12 years of age.
  Interventions: Device: iotaSOFT Insertion System

INTERVENTIONS:
Device: iotaSOFT Insertion System — robotic assistive technology for cochlear implant electrode insertion

SUMMARY:
Prospective, non-randomized, open-label study to evaluate the safety and efficacy of the iotaSOFT Insertion System when used to assist electrode array insertion during cochlear implant surgery in a pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for unilateral or bilateral cochlear implantation according to indications for use with FDA approved cochlear implant devices
* Age 9 months to less than 12 years old at the time of CI surgery
* Willingness to participate in the study and able to comply with the follow-up visit requirements

Exclusion Criteria:

* Prior cochlear implantation in the ear to be implanted
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array or present an increased risk of aberrant insertion
* Craniofacial abnormality, temporal squamosal skull thickness less than 3mm, major cochlear lesions, or cochlear malformations
* Deafness due to lesions of the acoustic nerve or central auditory pathway
* Diagnosis of auditory neuropathy.
* Active middle-ear infection or tympanic membrane perforation in the presence of active middle-ear disease
* Absence of cochlear development
* Additional medical concerns that would prevent participation in evaluations as determined by the investigator
* Planned or current participation in a clinical study of an investigational device or drug

Ages: 9 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Safety related to adverse events | 30 days following surgery
  Evaluation of iotaSOFT related adverse events and serious adverse events through 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Laura Chenier, Study Director — iotaMotion, Inc.
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Texas Childrens Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided